CLINICAL TRIAL: NCT01017822
Title: A Phase I/II Study of Induction Conatumumab and Gemcitabine, Followed by Conatumumab, Capecitabine and 3-D Conformal Radiation Therapy (3D-CRT) With Subsequent Maintenance Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Conatumumab, Gemcitabine Hydrochloride, Capecitabine, and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to study agent availability.
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0932; CDR0000659527
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — conatumumab; Capecitabine; Gemcitabine; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: conatumumab
Drug: capecitabine
Drug: gemcitabine hydrochloride
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as conatumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as gemcitabine hydrochloride and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy may uses high energy x-rays to kill tumor cells. Giving conatumumab together with gemcitabine hydrochloride, capecitabine, and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of conatumumab when given together with gemcitabine hydrochloride, capecitabine, and radiation therapy and to see how well they work in treating patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the maximum tolerated dose of conatumumab up to a target dose of 10 mg/kg given concurrently with capecitabine and radiotherapy following induction therapy comprising conatumumab and gemcitabine hydrochloride in patients with locally advanced pancreatic cancer. (Phase I)
* To evaluate the overall survival of patients treated with this regimen. (Phase II)

Secondary

* To evaluate the safety profile in patients treated with this regimen. (Phase I and II)
* To evaluate the progression-free survival of patients treated with this regimen. (Phase II)
* To evaluate the primary tumor response rate in patients treated with this regimen. (Phase II)
* To generate translational research hypotheses. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of conatumumab, followed by a phase II study.

* Induction therapy: Patients receive conatumumab IV over 30-60 minutes on days 1 and 15 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses.
* Conatumumab and chemoradiotherapy: Beginning 14-42 days after the last course of induction therapy, patients undergo 3-dimensional radiotherapy once daily, 5 days a week, for 5½ weeks (28 treatments). Patients also receive conatumumab IV over 30-60 minutes on days 1, 15, and 29 and oral capecitabine twice daily, 5 days a week, for 5½ weeks.
* Maintenance therapy: Beginning 28-56 days after completion of chemoradiotherapy, patients receive conatumumab IV over 30-60 minutes on days 1 and 15 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced disease
  * With and without regional adenopathy
* Unresectable disease based on institutional standardized criteria of unresectability OR medically inoperable
* No distant metastatic disease, second malignancy, or peritoneal seeding

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention allowed)
* Serum creatinine ≤ 1.5 mg/dL
* ALT or AST < 3 times upper limit of normal (ULN)
* Total bilirubin < 3.0 mg/dL
* Alkaline phosphatase < 3 times ULN
* Amylase ≤ 2 times ULN
* Lipase ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after the last study drug administration (for women) or for ≥ 6 months after the last study drug administration (for men)
* Able to swallow oral medications
* No other invasive malignancy within the past 2 years, except for nonmelanomatous skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No severe, active co-morbidity, including any of the following:

  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
  * Transmural myocardial infarction within the past 3 months
  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Any other cardiac condition that, in the opinion of the treating physician, would make study treatment unreasonably hazardous for the patient
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function
  * Any unresolved bowel or bile duct obstruction
  * Major resection of the stomach or small bowel that could affect the absorption of capecitabine
  * AIDS based upon current CDC definition

    * HIV testing is not required for study entry
* No prior allergic reaction to capecitabine or gemcitabine hydrochloride

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* No prior treatment with TRAIL-receptor agonists
* No prior systemic chemotherapy for pancreatic cancer
* More than 2 years since prior chemotherapy for malignancies other than pancreatic cancer
* More than 28 days since prior major surgery (e.g., biliary or gastric bypass)

  * Insertion of a vascular access device, exploratory laparotomy, or laparoscopy are not considered major surgery
* No concurrent intensity-modulated radiotherapy
* No other concurrent chemotherapy
* No other concurrent monoclonal antibody therapy
* No concurrent sorivudine, brivudine A, or cimetidine
* No concurrent participation in another clinical trial
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided INR is monitored

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Phase I)
Overall survival (Phase II)

SECONDARY OUTCOMES:
Adverse events (Phase I and II)
Progression-free survival (Phase II)
Response rate (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Crane, MD, Principal Investigator — M.D. Anderson Cancer Center